CLINICAL TRIAL: NCT05239845
Title: Evaluating the Effects of Prebiotic-based Interventions on Sleep, the Gut Microbiome, Cognition, Immune Function and Stress Following 56 Days Consumption in Healthy Volunteers
Brief Title: Evaluating the Effects of Prebiotics on Sleep, the Gut Microbiome, Cognition, Immune Function and Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Reckitt Benckiser Group PLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 35654
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Sleep
Keywords: Gut Microbiome; Stress; Immune Function; Cognition
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Investigational Supplement 1 (INV-1) (Active Comparator): The total daily supplement to be consumed by participants is 33.0 g. This will be administered as 2 separate doses mixed with water, a 16.5 g dose (two 8.25 g sachets) to be consumed in the morning (AM dose) and a 16.5 g dose (two 8.25 g sachets) to be consumed in the evening (PM dose). Supplementation will last 56 days.
  Interventions: Dietary Supplement: Prebiotic
- Investigational Supplement 1 (INV-2) (Active Comparator): The total daily supplement to be consumed by participants is 33.0 g. This will be administered as 2 separate doses mixed with water, a 16.5 g dose (two 8.25 g sachets) to be consumed in the morning (AM dose) and a 16.5 g dose (two 8.25 g sachets) to be consumed in the evening (PM dose). Supplementation will last 56 days.
  Interventions: Dietary Supplement: Prebiotic
- Investigational Supplement 1 (INV-3) (Active Comparator): The total daily supplement to be consumed by participants is 33.0 g. This will be administered as 2 separate doses mixed with water, a 16.5 g dose (two 8.25 g sachets) to be consumed in the morning (AM dose) and a 16.5 g dose (two 8.25 g sachets) to be consumed in the evening (PM dose). Supplementation will last 56 days.
  Interventions: Dietary Supplement: Prebiotic
- Control (Placebo Comparator): The total daily supplement to be consumed by participants is 33.0 g. This will be administered as 2 separate doses mixed with water, a 16.5 g dose (two 8.25 g sachets) to be consumed in the morning (AM dose) and a 16.5 g dose (two 8.25 g sachets) to be consumed in the evening (PM dose). Supplementation will last 56 days.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Prebiotic — The bioactive ingredients used in this study include bovine milk fat globule membrane (MFGM), bovine lactoferrin and a prebiotic blend of polydextrose and galactooligosaccharides (PDX/GOS).
  Arms: Investigational Supplement 1 (INV-1); Investigational Supplement 1 (INV-2); Investigational Supplement 1 (INV-3)
Other: Control — Maltodextrin
  Arms: Control

SUMMARY:
The aim of the proposed randomised, double-blind, controlled, parallel groups trial is to assess the sleep, gut microbiome, cognitive, immune and stress effects of 56 days administration of three formulations of a prebiotic-based intervention, in comparison to a placebo control, in a cohort of healthy adults reporting poor sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health.
* Have a stable sleep/wake schedule (bedtime between 9pm and 1am and wake time between 6am and 10am at least 5 nights per week)
* Aged 25 to 60 years at the time of randomisation
* Fluent in English
* Identify as a 'poor sleeper' as defined subjectively (i.e. poor sleep quality, unrefreshing sleep) and a total score of >5 on the Pittsburgh Sleep Quality Index (PSQI).

Exclusion Criteria:

* Member of own household currently participating in this trial
* Evidence of current or recent sleep disorders (e.g. sleep apnoea, insomnia, circadian rhythm disorders), taking any medication which exerts sedative effects, affects the CNS and/or sleep, or be currently unwell with any illness that affects sleep (i.e. disorders of the CNS). An initial screening for sleep disorders will be conducted using the Sleep Disorders Symptom Checklist-25 (SDS-CL; Klingman et al., 2017). If a participant reports positively to any of the 25 questions in terms of being affected for three nights per week, or more, this will be followed up using a clinical interview according to the International Classification of Sleep Disorders (ICSD-3) to exclude on the basis of a sleep disorder
* History of seizures or epilepsy
* Shift working or have a history of shift work within the previous six months
* Currently, or within the previous 8 weeks, consuming any prebiotic or probiotic products/supplements (including specifically oligosaccharides)
* Participation in any other intervention research trials
* Sleeping at a location other than their usual residence more than two nights per week during participation
* Travel across multiple time zones within the last three months or have planned travel across multiple time zones during the study
* Current or recent mood disturbances or Axis I disorders
* Current misuse of alcohol and/or drugs
* Current smoker
* Recent (within the last 12 weeks) infection and/or use of antibiotic medication
* Pregnant, seeking to become pregnant or lactating
* Those using (including within the last 2 weeks) proton-pump inhibitors
* Milk allergy

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lab-recorded polysomnography- Sleep Quality | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  percentage of time in staged sleep from total sleep recorded time

SECONDARY OUTCOMES:
Lab-recorded polysomnography- Sleep onset latency | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  minutes taken from intention to sleep to first epoch of any stage of sleep
Lab-recorded polysomnography- Total sleep time | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  minutes of staged sleep over entire sleep duration period
Lab-recorded polysomnography- Number of awakenings | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  number of <15 second bouts of Wake surrounded, at both ends, by any sleep stage
Lab-recorded polysomnography- Wake after sleep onset | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  cumulative minutes of scored Wake during entire sleep duration following sleep initiation
Lab-recorded polysomnography- Time spent in stages of rapid eye movement (REM) and non-REM sleep | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  percentage of time spent in REM, N1, N2, N3
Lab-recorded polysomnography- REM Rebound | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  length, frequency and depth of REM sleep
Lab-recorded polysomnography- Sleep microstructure | Change from protocol days 2 and 3 (baseline) and 59 and 60 following 56 days of supplement consumption
  including k-complexes - >.0.5 secs. negative then positive wave and fast/slow sleep spindles - >.0.5 secs. sinusoidal waves 11-16Hz
Actigraphy - Sleep onset latency | Change from baseline following 56 days of supplement consumption
  recorded minutes taken from intention to sleep to sleep initiation
Actigraphy - Total sleep time | Change from baseline following 56 days of supplement consumption
  recorded minutes asleep over entire sleep period
Actigraphy - Number of awakenings | Change from baseline following 56 days of supplement consumption
  recorded number of awakenings during entire sleep period
Actigraphy - Wake after sleep onset (WASO) | Change from baseline following 56 days of supplement consumption
  recorded minutes awake during the entire sleep period following sleep onset
Actigraphy - Sleep efficiency | Change from baseline following 56 days of supplement consumption
  ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed (percentage)
Blood Pressure and Heart Rate (BP/HR) | Change from baseline following 56 days of supplement consumption
  Measured using a fully automatic oscillometric device
Body Mass Index (BMI) | Change from baseline following 56 days of supplement consumption
  calculated using standard formula: weight (kg) / [height (m)]2
Waist-to-Hip Ratio (WHR) | Change from baseline following 56 days of supplement consumption
  WHR will be calculated by dividing waist circumference by hip circumference.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline following 56 days of supplement consumption
  Pittsburgh Sleep Quality Index (PSQI): Total Score. The PSQI is a validated self-rating instrument assessing aspects of sleep quality.Minimum score 0 (better); maximum score 21 (worse) < or = 5 associated with good sleep quality; > 5 associated with poor sleep quality.
Profile of Mood States (POMS) | Change from baseline following 56 days of supplement consumption
  Profile of Mood States (POMS): Mood scores. The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. 65 adjectives rated on 5-point scale 0= not at all; 1=a little; 2=moderately; 3=quite a bit; 4=extremely. Factor analysis: 6 subscales tension-anxiety (9 items, score range: 0-36) depression (15 items, range 0-60) anger-hostility (12 items, range 0-48) vigor-activity (8 items, range 0-32) fatigue (7 items, range 0-28) confusion-bewilderment (7 items, range 0-28) Total mood disturbance (TMD): (range 0-200)
Depression, Anxiety and Stress Scale - 21 Items (DASS-21) | Change from baseline following 56 days of supplement consumption
  A 21-item measure of mood over the previous week (each item is rated on scale from 0-3). Scoring creates 3 component scores: depression, anxiety and stress (each on a scale of 0-21) with higher scores indicating higher symptomology. Cut-off scores, according to each set of symptoms, are available (normal, mild, moderate, severe and extremely severe) or total scores can be derived by multiplying the sum of all three component scores by 2.
State-Trait Anxiety Inventory (STAI) | Change from baseline following 56 days of supplement consumption
  A 40-item measure of current and general anxiety levels. Each item is rated on a scale from 1-4. Scoring creates two components: state anxiety (20 items) and trait anxiety (20 items), with a range for each between 20-80. Following transformation through reversed coding, higher scores indicate higher levels of anxiety.
Work Productivity and Activity Impairment questionnaire (WPAI) | Change from baseline following 56 days of supplement consumption
  A 6-item measure of the impact of an individual's health on their work over the previous week. There are 4 component scores: presenteeism, activity impairment, absenteeism and overall work productivity. All items have varying response formats and higher scores indicate more impairment in each domain. Overall scores can also be summed and multiplied by 100 for an overall impairment index.
12-Item Short Form Survey (SF-12) | Change from baseline following 56 days of supplement consumption
  A 12-item measure of current perceptions of health status. All items have varying response formats and result in 8 component scores: 1) Limitations in physical activities because of health problems, 2) Limitations in social activities because of physical or emotional problems, 3) Limitations in usual role activities because of physical health problems, 4) Bodily pain, 5) General mental health (psychological distress and well-being), 6) Limitations in usual role activities because of emotional problems, 7) Vitality (energy and fatigue) and 8) General health perceptions.
Perceived Stress Scale (PSS | Change from baseline following 56 days of supplement consumption
  Perceived Stress Scale (PSS): Total Score. The PSS is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances.Participants rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56 higher scores indicate greater perceived stress
Gastrointestinal symptoms questionnaire | Change from baseline following 56 days of supplement consumption
  This in-house developed questionnaire is to be completed at the start and end of the trial, during the baseline and chronic lab visits respectively. When completing the assessment, participants will answer in relation to their experiences in the previous 7 days. The questionnaire asks 11 questions, plus a 12th open-ended question, about gastrointestinal experiences, with 5 possible ratings; 'not at all' (score of 0), 'A little' (score of 1), 'a moderate amount' (score of 2), 'quite a lot' (score of 3) and 'a severe amount' (score of 4). Scores can range between 0-44 with a higher score indicating a more negative experience of symptoms
Sleep Diary -Total Sleep Time | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual reports being asleep during the night between initiation and termination of sleep, accounting for nocturnal wake periods
Sleep Diary -Time in bed | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual reports being in bed intending to sleep
Sleep Diary -Sleep Latency | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual felt it took them to fall asleep after intending to sleep
Sleep Diary -Number of Awakenings | Change from baseline following 56 days of supplement consumption
  number of perceived awakenings over the sleep period
Sleep Diary - Wake After Sleep Onset (WASO) | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual reports being awake during the night after sleep initiation
Sleep Diary - Sleep Efficiency | Change from baseline following 56 days of supplement consumption
  Total Sleep Time divided by Time in Bed x 100, expressed as a percentage
Sleep Diary - Sleep Quality | Change from baseline following 56 days of supplement consumption
  4 items (each scored on a 0-4 scale) covering nocturnal physical and psychological tension, sleep enjoyment and feelings of restedness. Items can be summed (range 0-16) with higher scores indicating poorer sleep quality.
Dietary assessment- Intake24 | Change from baseline following 56 days of supplement consumption
  The Intake 24 measure (https://intake24.co.uk/) will assess participants dietary recall over the previous 24 hour period. The generated results provide an indication of overall calorie intake as well as fibre, sugar, calcium, total fat, saturated fat, vitamin C, iron, folate, fruit and vegetable and red meat intake.
Perceived sleep quality (VAS) | Change from baseline following 56 days of supplement consumption
  Assessed weekly via numerical rating scales. This will generate individual scores of 0-4 (0= 'Extremely poor' to 4= 'Extremely good')
Subjective Stress (VAS) | Change from baseline following 56 days of supplement consumption
  Assessed weekly via numerical rating scales. This will generate individual scores of 0-4 (0= 'Extremely poor' to 4= 'Extremely good')
Subjective mood (VAS) | Change from baseline following 56 days of supplement consumption
  Assessed weekly via numerical rating scales. This will generate individual scores of 0-4 (0= 'Extremely poor' to 4= 'Extremely good')
Subjective productivity (VAS) | Change from baseline following 56 days of supplement consumption
  Assessed weekly via numerical rating scales. This will generate individual scores of 0-4 (0= 'Extremely poor' to 4= 'Extremely good')
COMPASS global performance measures | Change from baseline following 56 days of supplement consumption
  Speed of performance, and accuracy of performance measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Cognitive domain factor score | Change from baseline following 56 days of supplement consumption
  Speed of attention, accuracy of attention, speed of memory, accuracy of working memory, and accuracy of episodic memory measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Cognitive Function under stressful conditions | Change from baseline following 56 days of supplement consumption
  Cognitive performance (multi tasking using Serial Subtractions (3s, 7s, 17s) and tracking simultaneously) during acute stress as a consequence of theOBSERVED MULTITASKING STRESSOR (OMS)
Changes in subjective stress; as assessed by the 'state, trait anxiety inventory' (STAI) | Change from baseline following 56 days of supplement consumption
  Subjective stress will be measured via the state, trait anxiety inventory before and after each completion of the observed multitasking stressor (OMS)
Changes in objective stress; as assessed by salivary cortisol levels | Change from baseline following 56 days of supplement consumption
  Saliva samples will be taken from participants before and after each completion of the observed multitasking stressor (OMS) and the change in salivary cortisol levels between pre- and post-OMS
Changes in objective stress; as assessed by salivary alpha-amylase levels | Change from baseline following 56 days of supplement consumption
  Saliva samples will be taken from participants before and after each completion of the observed multitasking stressor (OMS) and the change in salivary cortisol levels between pre- and post-OMS
Changes in objective stress; as assessed by galvanic skin response (GSR) | Change from baseline following 56 days of supplement consumption
  Galvanic skin response (GSR) will be recorded throughout the observed multitasking stressor (OMS)
Changes in objective stress; as assessed by heart rate (HR) | Change from baseline following 56 days of supplement consumption
  Heart rate (HR) will be recorded throughout the observed multitasking stressor (OMS)
Gut microbiome assessments (gut bacterial profile) | Change from baseline following 56 days of supplement consumption
  Assessed via analysis of self collected stool samples at baseline, during active supplementation and after 56 days of supplementation.
Immunological marker Assessment -Blood | Change from baseline following 56 days of supplement consumption
  Immune function (identification of blood biomarkers of immune function in samples collected at baseline and chronic lab visits)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ellis, PhD, Principal Investigator — Northumbria University
Locations (2):
- United Kingdom (2):
  - Northumbria Sleep Research, Northumbria University, Newcastle
  - Northumbria University, Newcastle

IPD SHARING:
Plan to Share IPD: No